CLINICAL TRIAL: NCT01562808
Title: The Relationship Between D2 Occupancy and Change in Frontal Metabolism and Working Memory Induced by Aripiprazole
Brief Title: Change in Brain Metabolism and Cognitive Function by Aripiprazole
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jun Soo Kwon, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: A070001
Record Dates: First submitted 2012-03-22; First posted 2012-03-26 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Antipsychotics; Cognition; Brain Metabolism; Dopamine Receptor Occupancy
MeSH Terms: interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Aripiprazole — single oral administration of aripiprazole

SUMMARY:
Dopamine receptor occupancy and brain metabolism were measured using positron emission tomography after the administration of aripiprazole. Working memory performance was also measured using N-back task.

The investigators explored the relationship between changes in brain metabolism and working memory performance.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers
* right-handed

Exclusion Criteria:

* any significant abnormality on routine lab
* any psychiatric disease

Ages: 19 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2009-01; Primary Completion 2010-05 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Reaction time of correct response in N-back task | 48 hrs after the administration of aripiprazole

CONTACTS AND LOCATIONS:
Overall Officials: Jun Soo Kwon, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea